CLINICAL TRIAL: NCT01423305
Title: Effect of Charcoal on Gastrointestinal Absorption of Budesonide and Formoterol
Brief Title: Phase I Pharmacokinetic Study (BF-BLOCK)
Acronym: BF-BLOCK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3103008
Record Dates: First submitted 2011-08-23; First posted 2011-08-25 (Estimated); Last update posted 2011-10-21 (Estimated); Status verified 2011-10

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide; Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Experimental): Budesonide/formoterol capsule (Orion Pharma) for oral administration.
  Interventions: Drug: Budesonide/formoterol capsule.
- Treatment B (Experimental): Budesonide/formoterol capsule (Orion Pharma) for oral administration.
  Interventions: Drug: Budesonide/formoterol capsule for oral adm.

INTERVENTIONS:
Drug: Budesonide/formoterol capsule. — Oral administration with concomitant charcoal.
  Arms: Treatment A
Drug: Budesonide/formoterol capsule for oral adm. — Oral administration without concomitant charcoal.
  Arms: Treatment B

SUMMARY:
The objective of the study is to assess if charcoal prevents the absorption of budesonide and formoterol via GI track. The assessment will be based on comparing the pharmacokinetic parameter area under the concentration-time curve.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females aged 18-60 years.
2. Normal weight at least 50 kg.

Exclusion Criteria:

1. Evidence of a clinically significant cardiovascular, renal, hepatic, haematological, gastrointestinal, pulmonary, metabolic-endocrine, neurological or psychiatric disease.
2. Any clinically significant abnormal laboratory value or physical finding that may interfere with the interpretation of study results or constitute a health risk for the subject if he/she takes part in the study.
3. Any condition requiring concomitant treatment (including vitamins and herbal products) or likely to need any concomitant treatment during the study.
4. Known hypersensitivity to the active substance(s) or the excipients of the drug.
5. Pregnant or lactating females.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
The evaluation of primary pharmacokinetic variable AUCt | 4 weeks
  The evaluation of primary pharmacokinetic variable AUCt of this study will be based on statistical methods appropriate for crossover design.

SECONDARY OUTCOMES:
Pharmacokinetic variables | 4 weeks
  Cmax
Pharmacokinetic variable | 4 weeks
  tmax

CONTACTS AND LOCATIONS:
Overall Officials: Mika Scheinin, M.D.Ph.D, Principal Investigator — Clinical Research Services Turku Finland
Locations (1):
- Clinical Reseach Services Turku (CRST), Turku, Finland